CLINICAL TRIAL: NCT04191031
Title: A Multicenter, Double-blind, Randomized, Sham-controlled Study Assessing Opioid Utilization, Postoperative Pain and Function in Subjects Undergoing Total Knee Arthroplasty Treated With Presurgical Iovera®° or Sham Iovera®° Cryoneurolysis and Postsurgical Multimodal Pain Regimen
Brief Title: Study to Evaluate Iovera®° in Adult Patients Undergoing Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: One of the pre-determined criteria for efficacy analysis in the interim analysis SAP for stopping the study was met.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOV-401
Record Dates: First submitted 2019-11-26; First posted 2019-12-09 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Post-Operative Pain Management
Keywords: Total Knee Arthroplasty; Osteoarthritis; Iovera
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Superficial Genicular Nerves (Experimental): Subjects will receive iovera° cryoneurolysis treatment of superficial genicular nerves (anterior femoral cutaneous nerve [AFCN] and infrapatellar branches of the saphenous nerve [ISN]) of the target knee
  Interventions: Device: ioveraº
- Sham Comparator (Sham Comparator): Subjects will receive sham iovera° treatment of superficial genicular nerves (AFCN and ISN) of the target knee
  Interventions: Device: ioveraº sham

INTERVENTIONS:
Device: ioveraº — Cryoneurolysis
  Arms: Superficial Genicular Nerves
Device: ioveraº sham — ioveraº sham
  Arms: Sham Comparator

SUMMARY:
Primary objective: The primary objective of this study is to evaluate postsurgical pain control, after presurgical iovera° treatment plus EXPAREL® and standardized multimodal therapy compared with presurgical sham iovera° treatment plus EXPAREL and standardized multimodal therapy in subjects undergoing primary unilateral total knee arthroplasty (TKA).

Secondary objectives: The secondary objectives of this study are to compare postsurgical pain control or postsurgical total opioid consumption, opioid-free status, physical function, sleep quality, and safety of presurgical iovera° treatment plus EXPAREL and standardized multimodal therapy with presurgical sham iovera° treatment plus EXPAREL and standardized multimodal therapy, in subjects undergoing primary unilateral TKA

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, sham-controlled study in adult subjects undergoing TKA. Approximately 200 subjects are planned for enrollment and will be randomized 1:1 to receive presurgical ioveraº treatment or sham ioveraº treatment. An unblinded interim analysis will be performed when approximately 60 randomized and treated subjects have completed the Day 30 assessments. Based on the results of the interim analysis, sample size re-estimation will be performed and one of the following will occur: (1) the study will proceed to the final analysis without additional interim analysis, (2) the study will proceed to the second interim analysis once a defined number of additional subjects have completed Day 30 assessments, at which time, the study may be stopped for success or futility or proceed to the final analysis (3) the study will be stopped for futility. The detailed decision rules are defined in response to the interim analysis statistical analysis plan (IA SAP).

This study is designed to investigate whether presurgical iovera° cryoneurolysis treatment leads to less postsurgical opioid consumption, decreased pain after surgery, improved function, and improved postsurgical outcomes compared with subjects who undergo presurgical sham iovera° treatment. All subjects will receive postsurgical multimodal pain medications and intraoperative local infiltration with EXPAREL (bupivacaine liposome injectable suspension).

Subjects may be screened within 60 days prior to TKA. No procedures other than the site's standard of care will be performed before signed informed consent is obtained. When screening test results are received and the subject is deemed eligible for the study, the subject will be notified that he or she can be enrolled in the study.

Subjects may be rescreened upon sponsor approval for administrative reasons.

Randomization to treatment groups and treatment with the iovera° system according to the randomization assignment will be performed prior to TKA. The treatment groups are:

* Group 1: subjects will receive iovera° cryoneurolysis treatment of superficial genicular nerves of the target knee
* Group 2: subjects will receive sham iovera° treatment of superficial genicular nerves of the target knee

At the subsequent TKA, all subjects in both groups will receive intraoperative local infiltration with EXPAREL and postsurgical multimodal pain medications.

After discharge, subjects will be followed for 90 days. Subjects will be assessed for safety, efficacy, and health outcomes parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 22 years of age at screening.
2. Scheduled to undergo primary, unilateral, tricompartmental TKA under spinal anesthesia.
3. Primary indication for TKA is degenerative osteoarthritis of the knee.
4. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
5. Anticipation of discharge to home after inpatient acute postsurgical phase based on age, comorbidities, home environment, social support, and the judgment of the Investigator.
6. Females of childbearing potential must have a negative pregnancy test result prior to enrollment and agree to use a highly effective method of birth control during the study. A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year). Post-menopausal or surgically sterile females would not require a pregnancy test.
7. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. History of prior contralateral TKA within 6 months or open knee surgery on the knee being considered for TKA. Prior arthroscopy is permitted.
2. Planned concurrent surgical procedure (e.g., bilateral TKA) or planned additional surgery within 90 days of study surgery.
3. Undergoing unicompartmental TKA or revision TKA.
4. Concurrent painful physical condition that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to the knee surgery and which may confound the postsurgical assessments (e.g., significant pain from other joints including the non-index knee joint, chronic neuropathic pain, concurrent or prior contralateral TKA, concurrent foot surgery).
5. Comorbidity that, in the judgment of the Investigator, may affect the subject's ability to participate in the study and postsurgical rehabilitation.
6. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications (i.e., bupivacaine, lidocaine, acetaminophen, tranexamic acid, celecoxib, naproxen, meloxicam).
7. Use of any of the following medications within the times specified before TKA: long-acting and short-acting opioid medications within 6 weeks; or NSAIDs (except for low-dose aspirin used for cardioprotection) within 3 days or 5 elimination half-lives, whichever is longer.
8. Initiation of treatment with any of the following medications within 1 month prior to the screening visit or ongoing concomitant use if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, he or she must be on a stable dose for at least 1 month prior to screening visit.
9. Current use of systemic glucocorticosteroids within 1 month prior to screening in this study, intra-articular corticosteroid injections within 6 weeks, or Zilretta within 3 months.
10. History of coronary or vascular stent placed within the past 6 months (may be extended to 1 year if medically indicated per physician discretion).
11. Have been treated for a deep vein thrombosis, pulmonary embolism, myocardial infarction, or ischemic stroke within the past 6 months (may be extended to 1 year if medically indicated per physician discretion).
12. Any clotting disorder and/or use of an anticoagulant (e.g. warfarin, clopidogrel, etc.) within seven (7) days prior to administration of ioveraº treatment.
13. Rheumatoid or inflammatory arthritis.
14. History of severely impaired renal or hepatic function (in the judgment of the investigator).
15. Any neurologic or psychiatric disorder that might affect postsurgical pain or interfere with study assessments.
16. Malignancy in the last 2 years, per physician discretion.
17. History of misuse, abuse, or dependence on opioid analgesics, other prescription drugs, illicit drugs, or alcohol within the past 2 years.
18. Use of marijuana, including medical use, within 6 weeks prior to screening visit or continuation thereafter.
19. Body weight <50 kg (110 pounds) or a body mass index >40 kg/m2.
20. Previous iovera° treatment.
21. Greater than 15° malalignment (varus or valgus) on presurgical radiograph.
22. Prior surgery in the treatment areas that may have altered the anatomy of nerves intended to be treated with the ioveraº system or result in scar tissue in the treatment area.
23. Open and/or infected wounds at or near the treatment site.
24. Any other local skin condition at the treatment sites that in the Investigator's judgment would adversely affect treatment or outcomes.
25. History of cryoglobulinemia.
26. History of paroxysmal cold hemoglobinuria.
27. History of cold urticaria.
28. History of Raynaud's disease.
29. Administration of an investigational product within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to screening, or planned administration of another investigational product or procedure during the subject's participation in this study

Given the COVID-19 pandemic, the subject must be medically fit/cleared for surgery by the investigator. If there is a concern about a subject's recent or potential exposure to COVID-19, or if the subject is not medically fit/cleared for surgery due to suspected COVID-19 illness/symptoms (or other serious illness), the subject must be excluded per Exclusion criterion #5.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
NRS "worst pain" intensity scores from first pain assessment post-TKA (Day 1) to Day 30. | Day 1 to Day 30

SECONDARY OUTCOMES:
Change of KOOS scores (English version LK 1.0) from TKA Pre-Surgery visit to Day 30 visit post-TKA | Day -3 to Day 30
NRS "worst pain" intensity scores from first pain assessment post-TKA (Day 1) to Day 15, Day 42, and Day 90. | Day 1 to Day 90
NRS "average pain" intensity scores from first pain assessment post-TKA (Day 1) to Day 15, Day 30, Day 42, and Day 90 | Day 1 to Day 90
Change of NRS current pain intensity scores (pain "right now") from pre-treatment to post-treatment at the iovera/sham treatment visit | Day 1 to Day 90
Total postsurgical opioid consumption in oral morphine equivalents through Day 15, Day 30, Day 42, and Day 90 | Day 1 to Day 90
Percentage of subjects who are opioid free from post-TKA through Day 30 | Day 1 to Day 30
Change of KOOS scores from screening visit to each of the following visits: TKA Pre-Surgery, Day 15, Day 30, Day 42, and Day 90 | Day -3 to Day 90
Physical function (pain with 10 M walk, pain with passive range of motion (ROM) to 90° or 110° and active ROM maximum degrees of flexion) at the following visits: Day 15, Day 30, Day 42, and Day 90. | Day 15 to Day 90
Acute postoperative sleep quality by NRS daily through the first 7 days post TKA | Day 1 to Day 8
Change of extended postoperative sleep quality by PROMIS 8A scores from screening visit to each of the following visits: TKA Pre-Surgery, Day 15, Day 30, Day 42, and Day 90. | Screening to Day 90
NRS "worst pain" itensity scores from 72 hours post-TKA (Day 4) to Day 30 | Day 4 to Day 30
NRS "average pain" intensity scores from 72 hours post-TKA (Day 4) to Day 30 | Day 4 to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Gary Nevins, DC, Study Director — Pacira Pharmaceuticals, Inc
Locations (7):
- United States (7):
  - Sah Orthopaedic Associates at the Institute for Joint Restoration, Fremont, California
  - Lotus Clinical Research, Pasadena, California
  - Phoenix Clinical Research, Tamarac, Florida
  - Towson Orthopaedic Associates, Towson, Maryland
  - Northwell Health, New York, New York
  - First Surgical Hospital, Bellaire, Texas
  - Legent Orthopedic Hospital, Carrollton, Texas

IPD SHARING:
Plan to Share IPD: No